CLINICAL TRIAL: NCT04238689
Title: Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics and Pharmacodynamics of Monoclonal Antibody TB31F in Healthy Malaria-naïve Adults in the Netherlands
Brief Title: Safety, Tolerability, and Pharmacokinetics and Pharmacodynamics of TB31F
Acronym: TB31F
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: NL69779.091.19
Record Dates: First submitted 2019-12-23; First posted 2020-01-23 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2021-01

CONDITIONS: Malaria,Falciparum
Keywords: malaria; monoclonal antibody; falciparum; TB31F; transmission blocking; gametocyte
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Intervention Model Description: Five groups will receive a single dose of mAb TB31F administered intravenously (groups 1-4) or subcutaneously (group 5). Group 1 (n=5) will receive 0.1 mg/kg TB31F, group 2 (n=5) will receive 1 mg/kg TB31F, group 3 (n=5) will receive 3 mg/kg TB31F, group 4 (n=5) will receive 10 mg/kg mAb TB31F, and group 5 will receive 100mg TB31F. Twenty-five (n=25) subjects will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 - 0.1mg/kg TB31F (Experimental): 0.1 mg/kg of monoclonal antibody TB31F is administered intravenously to 5 subjects. Subjects will be observed for the occurrence of any adverse events. There will be a minimum of 48 hours between TB31F administration to each subsequent volunteer. Subjects will be followed-up for 84 days. Escalation to the next higher dosage group will be dependent upon no safety signals arising.
  Interventions: Biological: TB31F
- Group 2 - 1mg/kg TB31F (Experimental): 1 mg/kg of monoclonal antibody TB31F is administered intravenously to 5 subjects. TB31F administration will be staggered such that the first subject will be administered mAb TB31F and observed for the occurrence of any adverse events. The second subject will not receive their dose of TB31F sooner than 2 days after the first subject has received TB31F. The remaining three subjects will receive their TB31F dose no sooner than 2 days after the second subject has been administered TB31F, with at least a one hour interval in administration of TB31F between each subject. Subjects will be followed-up for 84 days. Escalation to the next higher dosage group will be dependent upon no safety signals arising.
  Interventions: Biological: TB31F
- Group 3 - 3mg/kg TB31F (Experimental): 3 mg/kg of monoclonal antibody TB31F is administered intravenously to 5 subjects. TB31F administration will be staggered such that the first subject will be administered mAb TB31F and observed for the occurrence of any adverse events. The second subject will not receive their dose of TB31F sooner than 2 days after the first subject has received TB31F. The remaining three subjects will receive their TB31F dose no sooner than 2 days after the second subject has been administered TB31F, with at least a one hour interval in administration of TB31F between each subject. Subjects will be followed-up for 84 days. Escalation to the next higher dosage group will be dependent upon no safety signals arising.
  Interventions: Biological: TB31F
- Group 4 - 10mg/kg TB31F (Experimental): 10 mg/kg of monoclonal antibody TB31F is administered intravenously to 5 subjects. TB31F administration will be staggered such that the first subject will be administered mAb TB31F and observed for the occurrence of any adverse events. The second subject will not receive their dose of TB31F sooner than 2 days after the first subject has received TB31F. The remaining three subjects will receive their TB31F dose no sooner than 2 days after the second subject has been administered TB31F, with at least a one hour interval in administration of TB31F between each subject. Subjects will be followed-up for 84 days.
  Interventions: Biological: TB31F
- Group 5 - 100mg TB31F (Experimental): 100mg of monoclonal antibody TB31F is administered subcutaneously to 5 subjects. TB31F administration will be staggered such that the first subject will be administered mAb TB31F and observed for the occurrence of any adverse events. The second subject will not receive their dose of TB31F sooner than 2 days after the first subject has received TB31F. The remaining three subjects will receive their TB31F dose no sooner than 2 days after the second subject has been administered TB31F, with at least a one hour interval in administration of TB31F between each subject. Subjects will be followed-up for 84 days.
  Interventions: Biological: TB31F

INTERVENTIONS:
Biological: TB31F — Monoclonal antibody

SUMMARY:
This phase 1 study aims to assess the safety and tolerability of monoclonal antibody TB31F administered intravenously or subcutaneously at escalating dose levels in healthy, malaria naïve, adults. This study will also evaluate the pharmacokinetics of TB31F and the functional activity of mAb TB31F in the standard membrane feeding assay.

DETAILED DESCRIPTION:
This phase 1 study aims to assess the safety and tolerability of monoclonal antibody (mAb) TB31F administered intravenously or subcutaneously in healthy, malaria naïve, adults at the Radboud University Medical Center (Radboudumc). Five groups will receive a single dose of mAb TB31F. Group 1 (n=5) will receive 0.1 mg/kg TB31F, Group 2 (n=5) will receive 1 mg/kg TB31F, group 3 (n=5) will receive 3 mg/kg TB31F, and group 4 (n=5) will receive 10 mg/kg mAb TB31F intravenously. Group 5 will receive 100mg TB31F subcutaneously. Twenty-five (n=25) subjects will be enrolled, as well as 1 reserve subject per group. Safety follow-up will be done at following times: baseline, end of infusion (EOI), 1, 3, 6 and 24 hours and 2, 7, 14, 21, 28, 56 and 84 days after administration. Extra follow-up visits at 4 and 10 days after administration for collection of serum/plasma for pharmacokinetic and pharmacodynamic measurements will be performed in group 5.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must sign written informed consent to participate in the trial.
2. Subject is able to understand planned study procedures and demonstrate comprehension of the protocol procedures and knowledge of study by passing a quiz (assessment of understanding).
3. In the opinion of the investigator, the subject can and will comply with the requirements of the protocol.
4. Subjects are available to attend all study visits and are reachable by phone throughout the entire study period from day -1 until day 84 (end of study).
5. The subject will remain within reasonable travelling distance from the study center from day -1 until day +7 after mAb TB31F infusion.
6. Subject is a male or non-pregnant and non-lactating female age ≥ 18 and ≤ 35 years and in good health at time of mAb infusion.
7. Subject agrees to their general practitioner (GP) being informed about participation in the study and agrees to sign a form to request the release by their GP, and medical specialist when necessary, of any relevant medical information concerning possible contra-indications for participation in the study to the investigator(s).
8. The subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period according to current Sanquin guidelines.
9. Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause. All subjects must agree to use continuous adequate contraception until 2 months after completion of the study. Female subjects must agree not to breastfeed from 30 days prior to mAb infusion until 2 months after completion of the study. Female subject must have a negative pregnancy test at the inclusion visit.

Exclusion Criteria:

1. Acute or chronic disease at time of TB31F administration, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests:

   1. Acute disease is defined as the presence of a moderate or severe illness with or without fever. Subjects with a minor illness on the day of TB31F administration will be (temporarily) excluded from participation, but may be re-evaluated for inclusion at a later date. Subjects with a positive SARS-CoV2 test at inclusion will be (temporarily) excluded from participation but may be re-evaluated for inclusion at a later date (following current Radboudumc guidelines).
   2. Fever is defined as an oral, axillary or tympanic temperature ≥ 38.0°C (100.4°F). The preferred route for recording temperature in this study will be oral.
   3. Any abnormal and clinically significant baseline laboratory screening tests of alanine aminotransferase, aspartate aminotransferase, creatinine, hemoglobin, platelet count or total white blood cell count, as defined in the protocol according to the FDA Toxicity Grading Scale for Healthy Adult and Adolescent Subjects Enrolled in Preventative Vaccine Clinical Trials.
2. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.
3. Chronic use of i) immunosuppressive drugs, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.
4. Positive urine toxicology test for cannabis, cocaine or amphetamines at screening or at inclusion.
5. Screening tests positive for Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV).
6. Use of any investigational or non-registered product (drug or vaccine) during the study period other than the study product.
7. Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
8. Prior receipt of an investigational antimalarial monoclonal antibody.
9. History of adverse reactions to monoclonal antibodies.
10. Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study mAb or planned administration during the study period.
11. Any history of malaria, positive serology for P. falciparum, or previous participation in any malaria (vaccine) study or Controlled Human Malaria Infection.
12. Body weight >= 115 kg
13. Being an employee or student of the department of Medical Microbiology or Medium Care of the Radboudumc, or a person otherwise related to the investigator other than a professional relationship for clinical trial purpose only.
14. History of drug or alcohol abuse interfering with normal functioning in the period of one year prior to study onset.
15. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew BB McCall, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] van der Boor SC, Smit MJ, van Beek SW, Ramjith J, Teelen K, van de Vegte-Bolmer M, van Gemert GJ, Pickkers P, Wu Y, Locke E, Lee SM, Aponte J, King CR, Birkett AJ, Miura K, Ayorinde MA, Sauerwein RW, Ter Heine R, Ockenhouse CF, Bousema T, Jore MM, McCall MBB. Safety, tolerability, and Plasmodium falciparum transmission-reducing activity of monoclonal antibody TB31F: a single-centre, open-label, first-in-human, dose-escalation, phase 1 trial in healthy malaria-naive adults. Lancet Infect Dis. 2022 Nov;22(11):1596-1605. doi: 10.1016/S1473-3099(22)00428-5. Epub 2022 Aug 10. PMID 35963275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 23 January 2020 - 8 December 2020 Recruitment location: Radboudumc Technology Center Clinical Studies
Groups:
- Group 1 - 0,1mg/kg TB31F: 0.1 mg/kg of monoclonal antibody TB31F is administered intravenously to 5 subjects. Subjects will be observed for the occurrence of any adverse events. There will be a minimum of 48 hours between TB31F administration to each subsequent volunteer. Subjects will be followed-up for 84 days. Escalation to the next higher dosage group will be dependent upon no safety signals arising.
  TB31F: Monoclonal antibody
Period: Overall Study
Arm/Group | Group 1 - 0,1mg/kg TB31F | Group 2 - 1mg/kg TB31F | Group 3 - 3mg/kg TB31F | Group 4 - 10mg/kg TB31F | Group 5 - 100mg TB31F
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - 0,1mg/kg TB31F | Group 2 - 1mg/kg TB31F | Group 3 - 3mg/kg TB31F | Group 4 - 10mg/kg TB31F | Group 5 - 100mg TB31F | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 25
Age, Continuous [Mean (Full Range); unit: years] | 22.0 [21.0 to 24.0] | 24.8 [22.0 to 26.0] | 26.8 [24.0 to 34.0] | 21.6 [19.0 to 25.0] | 22.2 [19.0 to 25.0] | 23.5 [19.0 to 34.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 4 | 1 | 13
  Male | 2 | 2 | 3 | 1 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 4 | 4 | 4 | 5 | 5 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Full Range); unit: kilograms] | 73.6 [60.4 to 84.8] | 75.5 [68.8 to 91.2] | 72.0 [53.0 to 86.0] | 71.5 [63.2 to 91.8] | 78.4 [63.0 to 93.0] | 74.2 [53.0 to 93.0]
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 24.3 [19.5 to 29.5] | 25.0 [22.0 to 27.8] | 23.4 [21.6 to 26.4] | 23.9 [21.7 to 29.0] | 23.9 [21.7 to 25.0] | 24.1 [19.5 to 29.5]

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Adverse Events After TB31F Administration
Description: * Number and severity of solicited local adverse events of all severities from first product administration through day 7;
  * Number and severity of solicited general adverse events and clinically significant hematological and biochemical laboratory abnormalities from first product administration through day 28;
  * Number and severity of unsolicited adverse events from first product administration through end of study;
  * Occurrence of serious adverse events from first product administration through end of study
Time Frame: Throughout study: solicited local adverse events (day 0 - day 7); solicited general adverse events and clinically significant laboratory abnormalities (day 0 - day 28); unsolicited adverse events (day 0 - day 84), serious adverse events (day 0 - day 84)
Population: Number of volunteers that experienced a grade 1, 2 or 3 local solicited, general solicited, unsolicited or laboratory adverse event per group.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - 0,1mg/kg TB31F | Group 2 - 1mg/kg TB31F | Group 3 - 3mg/kg TB31F | Group 4 - 10mg/kg TB31F | Group 5 - 100mg TB31F
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Participants
  Local Solicited Adverse Events: grade 1 | 0 | 1 | 1 | 0 | 4
  Local Solicited Adverse Events: grade 2 | 0 | 0 | 0 | 0 | 0
  Local Solicited Adverse Events: grade 3 | 0 | 0 | 0 | 0 | 0
  General Solicited Adverse Events: grade 1 | 4 | 3 | 1 | 5 | 2
  General Solicited Adverse Events: grade 2 | 3 | 0 | 0 | 1 | 0
  General Solicited Adverse Events: grade 3 | 0 | 0 | 0 | 0 | 0
  Unsolicited Solicited Adverse Events: grade 1 | 1 | 1 | 0 | 1 | 0
  Unsolicited Solicited Adverse Events: grade 2 | 1 | 0 | 0 | 0 | 0
  Unsolicited Solicited Adverse Events: grade 3 | 0 | 0 | 0 | 0 | 0
  Laboratory Adverse Events grade 1 | 1 | 1 | 0 | 0 | 2
  Laboratory Adverse Events grade 2 | 0 | 1 | 0 | 0 | 0
  Laboratory Adverse Events grade 3 | 0 | 0 | 0 | 0 | 0
  Laboratory Adverse Events where grade N/A, per protocol | 1 | 1 | 0 | 0 | 0
  Serious Adverse Event (SAE) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Serum Concentration of TB31F
Description: The serum concentration of TB31F will be measured in all subjects throughout the study (until day 84) by Pfs48/45 antigen ELISA.
Time Frame: All groups: 6 hours, 24 hours, 48 hours, day 7, day 14, day 21, day 28, day 56, day 84. Groups 1-4 only: end of infusion, 1 hour, 3 hours. Group 5 only: day 4 and day 10.
Population: Day 4 and day 10 were not measured for participants in groups 1 to 4, per protocol. Day 56 was not measured for group 1 participants due to COVID-19 pandemic-related restrictions.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 - 0,1mg/kg TB31F | Group 2 - 1mg/kg TB31F | Group 3 - 3mg/kg TB31F | Group 4 - 10mg/kg TB31F | Group 5 - 100mg TB31F
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4
ug/mL
  End of Infusion: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0
  End of Infusion | 2.59 (0.47) | 21.03 (3.34) | 79.54 (15.09) | 253.91 (51.27) |
  1 hour: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0
  1 hour | 2.80 (0.26) | 29.75 (11.11) | 69.77 (17.34) | 237.85 (45.91) |
  3 hours: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0
  3 hours | 2.84 (0.46) | 21.29 (3.65) | 75.28 (16.70) | 210.06 (56.72) |
  6 hours | 2.47 (0.27) | 19.30 (3.86) | 63.68 (15.15) | 165.45 (25.71) | 1.35 (0.64)
  24 hours | 2.17 (0.18) | 19.66 (3.37) | 56.51 (9.61) | 172.26 (69.10) | 4.08 (2.30)
  48 hours | 2.02 (0.15) | 15.28 (2.38) | 46.38 (8.61) | 139.56 (32.76) | 5.95 (3.29)
  Day 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Day 4 |  |  |  |  | 9.41 (4.15)
  Day 7 | 1.31 (0.09) | 9.65 (1.83) | 39.93 (5.61) | 118.03 (24.28) | 7.78 (3.30)
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Day 10 |  |  |  |  | 8.49 (3.28)
  Day 14 | 1.11 (0.16) | 7.14 (1.44) | 33.12 (0.55) | 91.61 (32.05) | 8.72 (4.90)
  Day 21 | 0.91 (0.11) | 8.07 (4.52) | 25.01 (4.17) | 67.87 (15.39) | 5.88 (2.18)
  Day 28 | 0.81 (0.11) | 4.99 (0.74) | 19.38 (3.51) | 69.55 (28.86) | 5.11 (1.92)
  Day 56: number analyzed (Participants) | 0 | 5 | 5 | 5 | 4
  Day 56 |  | 3.08 (0.52) | 9.52 (2.40) | 28.28 (6.78) | 2.86 (1.21)
  Day 84 | 0.30 (0.11) | 1.48 (0.43) | 4.88 (1.43) | 16.36 (4.62) | 1.77 (0.94)

3. Secondary Outcome: Pharmacodynamics/Functional Transmission-reducing Activity of TB31F
Description: Transmission-reducing activity (TRA) of serum TB31F will be assessed in all subjects throughout the study (until day 84) by standard membrane feeding assays (SMFA). TRA is expressed as the percentage reduction in oocysts in mosquitoes fed on gametocytes in the presence of participants' serum, compared to oocysts in mosquitoes fed on gametocytes in the presence of pooled naïve serum (control). Given the limited precision of low TRA estimates and the historical threshold value of >80% TRA to support clinical development of transmission-blocking vaccines, TRA >80% was pre-defined as the efficacy threshold of interest.
Time Frame: Groups 1 to 4: throughout study until day 84 (baseline, end of infusion, day 7, day 28, day 56, day 84). Group 5: baseline, day 2, day 4, day 7. day 10, day 14, day 28, day 56, day 84.
Population: Day 2, day 4, day 10, and day 14 were not measured for participants in groups 1 to 4, per protocol. For group 1 participants, analyses were not performed after end of infusion due to transmission reducing activity<80% at this timepoint.
Measure: Mean (Standard Deviation); unit: % Transmission Reducing Activity
Arm/Group | Group 1 - 0,1mg/kg TB31F | Group 2 - 1mg/kg TB31F | Group 3 - 3mg/kg TB31F | Group 4 - 10mg/kg TB31F | Group 5 - 100mg TB31F
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4
% Transmission Reducing Activity
  Pre-infusion | -23.52 (26.40) | 11.75 (25.15) | -45.24 (28.69) | -20.80 (36.94) | -24.89 (19.09)
  End of Infusion: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0
  End of Infusion | 46.88 (18.27) | 100.00 (0.00) | 99.91 (0.19) | 99.98 (0.05) |
  Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Day 2 |  |  |  |  | 96.40 (6.90)
  Day 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Day 4 |  |  |  |  | 99.69 (0.38)
  Day 7: number analyzed (Participants) | 0 | 5 | 5 | 5 | 4
  Day 7 |  | 99.71 (0.35) | 99.91 (0.12) | 100.00 (0.00) | 100.00 (0.00)
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Day 10 |  |  |  |  | 100.00 (0.00)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Day 14 |  |  |  |  | 99.39 (0.66)
  Day 28: number analyzed (Participants) | 0 | 5 | 5 | 5 | 4
  Day 28 |  | 95.41 (3.05) | 99.83 (0.28) | 99.87 (0.14) | 97.47 (4.03)
  Day 56: number analyzed (Participants) | 0 | 5 | 5 | 5 | 4
  Day 56 |  | 56.50 (30.80) | 96.09 (4.15) | 99.92 (0.08) | 78.67 (25.77)
  Day 84: number analyzed (Participants) | 0 | 5 | 5 | 5 | 4
  Day 84 |  | 18.87 (33.22) | 73.58 (27.74) | 99.73 (0.11) | 43.59 (57.13)

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | Group 1 - 0,1mg/kg TB31F | Group 2 - 1mg/kg TB31F | Group 3 - 3mg/kg TB31F | Group 4 - 10mg/kg TB31F | Group 5 - 100mg TB31F
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 4/5 | 2/5 | 5/5 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - 0,1mg/kg TB31F (N=5) | Group 2 - 1mg/kg TB31F (N=5) | Group 3 - 3mg/kg TB31F (N=5) | Group 4 - 10mg/kg TB31F (N=5) | Group 5 - 100mg TB31F (N=5)
Pain at site of injection (M79.68) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Redness at site of injection (L53.8) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling at site of injection (R22.9) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (R50.9) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (R51) (General disorders) | 1 (1) | 2 (4) | 0 (0) | 3 (7) | 0 (0)
Myalgia (M79.17) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (R53) (General disorders) | 5 (7) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Chills (R50.8) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (L98.9) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed feeling (F38) (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diahrrea (R19.4) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore Throat (J02.3) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach Ache (R10.4) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT04238689/Prot_001.pdf
  • Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT04238689/SAP_000.pdf